CLINICAL TRIAL: NCT04698473
Title: Comparison of Efficacy of Less Invasive Surfactant Treatment Under Nasal CPAP and Nasal IPPV in Premature Babies: CURLISPAP Study
Brief Title: Comparison of Efficacy of Less Invasive Surfactant Treatment Under Nasal CPAP and Nasal IPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hilal Ozkan, Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-AKD-138
Record Dates: First submitted 2020-12-15; First posted 2021-01-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: NCPAP; NIPPV; LISA
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCPAP (Active Comparator): Ventilator-derived NCPAP will be administered using binasal prongs. Standard Devices or infant flow-driver device. Initial NCPAP settings are: PEEP:6 cmH2O and FiO2: adjusted to keep preductal sPO2 between %90-94.
  Failure is defined as FiO2 requirement of >%50, capillary blood gas obtained at the 4th hour of therapy showing pH<7.20 or pCO2>60 cmH2O.
  Interventions: Other: NCPAP; Other: NIPPV
- NIPPV (Active Comparator): Ventilator-derived NIPPV will be administered using binasal prongs. Standard Devices or infant flow-driver device. Initial NIPPV settings are: PEEP:6 cmH2O, PIP: 15 cmH2O, Rate: 30-40/ bpm and FiO2: adjusted to keep preductal sPO2 between %90-94.
  Failure is defined as FiO2 requirement of >%50, capillary blood gas obtained at the 4th hour of therapy showing pH<7.20 or pCO2>60 cmH2O.
  Interventions: Other: NCPAP; Other: NIPPV

INTERVENTIONS:
Other: NCPAP — NCPAP infants will be randomized into two different non invasive ventilation groups
Other: NIPPV — NIPPV NCPAP infants will be randomized into two different non invasive ventilation groups

SUMMARY:
Non invasive ventilation is important in the care of preterm infants with respiratory failure, and surfactant treatment can be use with non invasive ventilation. However, there is no consensus on the best non-invasive ventilation mode for surfactant treatment in preterm infants.

Objective: To compare the effectiveness of nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (CPAP) in preterm infants ≤ 29 week gestational age.

DETAILED DESCRIPTION:
This CURLISPAP study was a multicenter, randomized controlled study at six level III neonatal intensive care units (NICUs) in Turkey. The protocol was approved by the ethics committee of each participating centre and Turkish Ministry of Health, Turkish Medicines and Medical Devices Agency.

Non invasive ventilated preterm infants with respiratory distress syndrome and gestational age from 241/7 weeks to 296/7 weeks were enrolled within 6 h of birth. Infants with major congenital malformations, need of mechanical ventiation, need of entubation in delivery room and lack of parental consent were excluded. Enrolled infants will randomize into two study groups (NIPPV group and CPAP group). The short binasal prongs will use as interface. For all the groups, if the fraction of inspired oxygen (FiO2) requirement is persistently higher than 0.30 target SpO2 90-94%.

For all groups Surfactant by "LISA" technique and with special catheter (LISAcath, Chiesi Pharmaceutics) of surfactant (Curosurf, Chiesi Pharmaceutics) 200 mg/kg.

The primary end-point, need of mechanical ventilation within 72 hours following surfactant treatment, will compared between the groups. Short and long-term neonatal outcomes will also evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 -29 week
* Clinical and radiological diagnosis of RDS
* Born in a hospital with a study center
* Spontaneous breathing
* Within the first 6 hours
* Non-invasive ventilation and FiO2 requirement >0.30
* Parental concent

Exclusion Criteria:

* Major congenital malformations
* Need of mechanical ventiation
* Need of entubation in delivery room
* Air weak syndrome
* No parental concent

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Treatment failure within 72 hours after randomization 72 hours after randomization | within 72 hours after randomization
  Need for invasive mechanical ventilation

SECONDARY OUTCOMES:
Rate of bronchopulmonary dysplasia | 36 weeks of postmenstrual age ]
  defined according to the NICHD definition

CONTACTS AND LOCATIONS:
Overall Officials: hilal ozkan, Study Director — Study director
Locations (1):
- Hilal Ozkan, Bursa, Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gopel W, Kribs A, Ziegler A, Laux R, Hoehn T, Wieg C, Siegel J, Avenarius S, von der Wense A, Vochem M, Groneck P, Weller U, Moller J, Hartel C, Haller S, Roth B, Herting E; German Neonatal Network. Avoidance of mechanical ventilation by surfactant treatment of spontaneously breathing preterm infants (AMV): an open-label, randomised, controlled trial. Lancet. 2011 Nov 5;378(9803):1627-34. doi: 10.1016/S0140-6736(11)60986-0. Epub 2011 Sep 29. PMID 21963186
- [Result] Lemyre B, Laughon M, Bose C, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD005384. doi: 10.1002/14651858.CD005384.pub2. PMID 27976361

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04698473/Prot_SAP_002.pdf